CLINICAL TRIAL: NCT04469049
Title: Mindfulness-based Cognitive Therapy for People With Parkinson's Disease and Caregivers
Brief Title: MBCT for People With Parkinson's Disease and Caregivers
Acronym: MBCT-PD-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Mount Zion Health Fund (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MZHF_20200962
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Parkinson Disease; Anxiety; Depression
Keywords: Parkinson's disease; Mindfulness-based intervention; Mindfulness-based cognitive therapy (MBCT)
MeSH Terms: conditions — Parkinson Disease; Anxiety Disorders; Depression | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: All participants will receive the MBCT intervention, however they will be separated in several distinct groups over time, due to MBCT protocol limitations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness-based cognitive therapy (MBCT) (Experimental): All participants will receive the MBCT intervention, consisting of 8 90-minute weekly group sessions.
  Interventions: Behavioral: Mindfulness-based cognitive therapy (MBCT)

INTERVENTIONS:
Behavioral: Mindfulness-based cognitive therapy (MBCT) — MBCT is an evidence-based psychotherapy which combines mindfulness skills with cognitive therapy strategies.

SUMMARY:
This study aims to explore the feasibility and effectiveness of mindfulness-based cognitive therapy (MBCT) in reducing anxiety and/or depressive symptoms in people with Parkinson's disease (PD) and caregivers of people with PD.

DETAILED DESCRIPTION:
An adapted MBCT intervention will be offered to people with Parkinson's disease (PD) and mild-to-moderate depression and/or anxiety, as well as caregivers of people with PD. Several 8-week long MBCT groups will be held between September 2020 and May 2021, based on the adapted protocol. The MBCT intervention will consist of 90-minute weekly groups focused on teaching mindfulness techniques and ways to recognize cognitive patterns that can increase anxiety and/or depression. Participants will be recruited from the community, according to the eligibility criteria detailed below. For all participants, the pre- and post-MBCT anxiety and/or depressive symptom severity and mindfulness levels (as measured with standardized, validated scales) will be compared, using a paired t-test. For caregivers, pre- and post-MBCT caregiver burden scores will be compared as well.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of Parkinson's disease (PD) or parkinsonism, established by a neurologist, or being a caregiver of a person with PD or parkinsonism
* Being able and willing to attend 8 weekly 90-minute online group sessions (5-6:30 pm PST)
* Mild-to-moderate anxiety: GAD-7 score ≤ 16
* Mild-to-moderate depression: PHQ-9 score ≤ 18

Exclusion Criteria:

* Severe anxiety: GAD-7 score > 16
* Moderately severe-to-severe depression: PHQ-9 score > 18
* Cognitive impairment: Montreal Cognitive Assessment (MoCA) score < 24
* Heavy alcohol or drug use
* Severe psychosis
* Active suicidal or homicidal ideation
* For people with PD: severe motor fluctuations (less than 2 hours "on" time per day)
* Pattern of engagement with health care that indicates low likelihood of completing an 8-week intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Change in anxiety symptom severity | From pre- to post-MBCT 8 weeks later
  Change in Generalized Anxiety Disorder-7 item score (for participants with anxiety). The scale score range is 0-21, with higher scores indicating more severe anxiety.
Change in depressive symptom severity | From pre- to post-MBCT 8 weeks later
  Change in Patient Health Questionnaire-9 score (for participants with depression). The scale score range is 0-27, with higher scores indicating more severe depression.

SECONDARY OUTCOMES:
Change in mindfulness levels | From pre- to post-MBCT 8 weeks later
  Change in 15 item-Five Facet Mindfulness Questionnaire score. The scale score range is 0-75, with higher scores indicating higher mindfulness levels.
Change in caregiver burden score (caregivers only) | From pre- to post-MBCT 8 weeks later
  Change in AMA Caregiver Self-Assessment Questionnaire score. The scale score range is 0-16, with higher scores indicating higher caregiver burden.

CONTACTS AND LOCATIONS:
Overall Officials: Andreea L. Seritan, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaudhuri KR, Healy DG, Schapira AH; National Institute for Clinical Excellence. Non-motor symptoms of Parkinson's disease: diagnosis and management. Lancet Neurol. 2006 Mar;5(3):235-45. doi: 10.1016/S1474-4422(06)70373-8. PMID 16488379
- [Background] Broen MP, Narayen NE, Kuijf ML, Dissanayaka NN, Leentjens AF. Prevalence of anxiety in Parkinson's disease: A systematic review and meta-analysis. Mov Disord. 2016 Aug;31(8):1125-33. doi: 10.1002/mds.26643. Epub 2016 Apr 29. PMID 27125963
- [Background] Reijnders JS, Ehrt U, Weber WE, Aarsland D, Leentjens AF. A systematic review of prevalence studies of depression in Parkinson's disease. Mov Disord. 2008 Jan 30;23(2):183-9; quiz 313. doi: 10.1002/mds.21803. PMID 17987654
- [Background] Martinez-Fernandez R, Schmitt E, Martinez-Martin P, Krack P. The hidden sister of motor fluctuations in Parkinson's disease: A review on nonmotor fluctuations. Mov Disord. 2016 Aug;31(8):1080-94. doi: 10.1002/mds.26731. Epub 2016 Jul 19. PMID 27431515
- [Background] Seritan AL, Ureste PJ, Duong T, Ostrem JL. Psychopharmacology for patients with Parkinson's disease and deep brain stimulation: Lessons learned in an academic center. Current Psychopharmacology 8(1):41-54, 2019 DOI: 10.2174/2211556007666180328142953
- [Background] Gotink RA, Chu P, Busschbach JJ, Benson H, Fricchione GL, Hunink MG. Standardised mindfulness-based interventions in healthcare: an overview of systematic reviews and meta-analyses of RCTs. PLoS One. 2015 Apr 16;10(4):e0124344. doi: 10.1371/journal.pone.0124344. eCollection 2015. PMID 25881019 (Retraction: PMID 30978236 PLoS One. 2019 Apr 12;14(4):e0215608)
- [Background] Cash TV, Ekouevi VS, Kilbourn C, Lageman SK. Pilot study of a mindfulness-based group intervention for individuals with Parkinson's disease and their caregivers. Mindfulness 7: 361-371, 2016
- [Background] Pickut B, Vanneste S, Hirsch MA, Van Hecke W, Kerckhofs E, Marien P, Parizel PM, Crosiers D, Cras P. Mindfulness Training among Individuals with Parkinson's Disease: Neurobehavioral Effects. Parkinsons Dis. 2015;2015:816404. doi: 10.1155/2015/816404. Epub 2015 May 26. PMID 26101690
- [Background] Dissanayaka NN, Idu Jion F, Pachana NA, O'Sullivan JD, Marsh R, Byrne GJ, Harnett P. Mindfulness for Motor and Nonmotor Dysfunctions in Parkinson's Disease. Parkinsons Dis. 2016;2016:7109052. doi: 10.1155/2016/7109052. Epub 2016 Apr 10. PMID 27144052
- [Background] Fitzpatrick L, Simpson J, Smith A. A qualitative analysis of mindfulness-based cognitive therapy (MBCT) in Parkinson's disease. Psychol Psychother. 2010 Jun;83(Pt 2):179-92. doi: 10.1348/147608309X471514. Epub 2009 Oct 19. PMID 19843353
- [Background] Rodgers SH, Schutze R, Gasson N, Anderson RA, Kane RT, Starkstein S, Morgan-Lowes K, Egan SJ. Modified Mindfulness-Based Cognitive Therapy for Depressive Symptoms in Parkinson's Disease: a Pilot Trial. Behav Cogn Psychother. 2019 Jul;47(4):446-461. doi: 10.1017/S135246581800070X. Epub 2019 Jan 18. PMID 30654854
- [Background] Teasdale JD, Segal ZV, Williams JM, Ridgeway VA, Soulsby JM, Lau MA. Prevention of relapse/recurrence in major depression by mindfulness-based cognitive therapy. J Consult Clin Psychol. 2000 Aug;68(4):615-23. doi: 10.1037//0022-006x.68.4.615. PMID 10965637
- [Background] Evans S, Ferrando S, Findler M, Stowell C, Smart C, Haglin D. Mindfulness-based cognitive therapy for generalized anxiety disorder. J Anxiety Disord. 2008 May;22(4):716-21. doi: 10.1016/j.janxdis.2007.07.005. Epub 2007 Jul 22. PMID 17765453
- [Background] Eisendrath SJ, Gillung E, Delucchi KL, Segal ZV, Nelson JC, McInnes LA, Mathalon DH, Feldman MD. A Randomized Controlled Trial of Mindfulness-Based Cognitive Therapy for Treatment-Resistant Depression. Psychother Psychosom. 2016;85(2):99-110. doi: 10.1159/000442260. Epub 2016 Jan 26. PMID 26808973
- [Derived] Seritan AL, Iosif AM, Prakash P, Wang SS, Eisendrath S. Online Mindfulness-Based Cognitive Therapy for People with Parkinson's Disease and Their Caregivers: a Pilot Study. J Technol Behav Sci. 2022;7(3):381-395. doi: 10.1007/s41347-022-00261-7. Epub 2022 May 2. PMID 35527798